CLINICAL TRIAL: NCT02517489
Title: Effects of Low-dose Corticosteroids on Survival of Severe Community-acquired Pneumonia
Brief Title: Community-Acquired Pneumonia : Evaluation of Corticosteroids
Acronym: CAPE_COD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PHRN14-PFD/CAPE COD
Record Dates: First submitted 2015-07-31; First posted 2015-08-07 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2023-01

CONDITIONS: Community Acquired Pneumonia
Keywords: Community-Acquired Pneumonia (CAP); Hydrocortisone; Corticosteroids; COronaVIrus Disease
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrocortisone (Experimental): Patients in the treatment group will receive intra-venous hydrocortisone (in addition to the standard treatment of severe Community-Acquired Pneumonia (CAP)
  Interventions: Drug: Hydrocortisone
- Placebo (Placebo Comparator): Patients of the control group will receive an intravenous placebo by intravenous route (in addition to the standard treatment of severe Community-Acquired Pneumonia (CAP)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydrocortisone — Hydrocortisone will be given in a double-blind fashion for 8 or 14 full days. The intravenous route will be used. The treatment course will include 4 or 7 days of full dose (200 mg/day by continuous infusion), 2 or 4 days of half dose (100 mg/day by continuous infusion), and 2 or 3 days of tapering dose (50 mg/day by continuous infusion). Duration of treatment is chosen upon patient initial improvement.
  Arms: Hydrocortisone
Drug: Placebo — Placebo will be given in a double-blind fashion for 8 or 14 full days. The intravenous route will be used. The treatment course will include 4 or 7 days of full dose (200 mg/day by continuous infusion), 2 or 4 days of half dose (100 mg/day by continuous infusion), and 2 or 3 days of tapering dose (50 mg/day by continuous infusion). Duration of treatment is chosen upon patient initial improvement.
  Arms: Placebo

SUMMARY:
Mortality of severe Community-Acquired Pneumonia (CAP) has not declined over time and is between 25 and 30% in sub-groups of patients. Corticosteroids (CTx) could down-regulate pulmonary and systemic inflammation, accelerate clinical resolution and decrease the rate of inflammation-associated systemic complications. Two recent meta-analyses suggest a positive effect on severe CAP day 28 survival when CTx are added to standard therapy. However they are based on only four trials gathering less than 300 patients, of which only one was positive. Recently published guidelines do not recommend CTx as part of CAP treatment. Therefore a well-powered trial appears necessary to test the hypothesis that CTx - and more specifically hydrocortisone - could improve day 28 survival of critically-ill patients with severe CAP, severity being assessed either on a Pulmonary Severity Index ≥ 130 (Fine class V) or by the use of mechanical ventilation or high-FiO2 high-flow oxygen therapy.

A phase-III multicenter add-on randomized controlled double-blind superiority trial assessing the efficacy of hydrocortisone vs. placebo on Day 28 all-causes mortality, in addition to antibiotics and supportive care, including the correction of hypoxemia.

Randomization will be stratified on: (i) centers; (ii) use of mechanical ventilation at the time of inclusion.

DETAILED DESCRIPTION:
Patients will receive state-of-the-art standard therapy for severe Community-Acquired Pneumonia (CAP), including antibiotics and supportive care. Correction of hypoxemia will use standard low-flow oxygen therapy, high-flow oxygen therapy, non-invasive-ventilation or invasive ventilation with endotracheal tube, as required. Patients in the treatment group will receive intra-venous hydrocortisone. Patients of the control group will receive an intravenous placebo by intravenous route at the same frequency.

Hydrocortisone or placebo will be given in a double-blind fashion for 8 or 14 full days. The intravenous route will be used. The treatment course will include 4 or 7 days of full dose (200 mg/day by continuous infusion), 2 or 4 days of half dose (100 mg/day by continuous infusion), and 2 or 3 days of tapering dose (50 mg/day by continuous infusion). Duration of treatment is chosen upon patient initial improvement.

A substantial amendment to the CAPE COD study has been submitted to the Competent Authorities in order to conduct a specific analysis on the sub-group of patients included with COVID19 (coronavirus disease 2019), in order to get a quick response in this specific population and in the context of an epidemic emergency.

The aim is to answer as quickly as possible a therapeutic question of major importance in the treatment of severe respiratory infections with CoV-2 SARS (severe acute respiratory syndrome coronavirus 2). Modifications made to the original study for patients with COVID (coronavirus disease) include some inclusion criteria, the primary endpoint, and secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients affiliated to social security scheme
* Admission to an Intensive Care Unit (ICU) or intermediate care unit participating to the trial
* Diagnosis of Community- Acquired Pneumonia (CAP) suggested by at least two of the following: cough, purulent sputum, chest pain and dyspnea
* Focal shadowing/infiltrate on chest X-ray or CT-scan
* Diagnosis of Community- Acquired Pneumonia (CAP) during the 48 hours post-hospital admission
* Study drug infusion initiated no longer than 24 hours post first severity criterion
* Severity defined by at least one of the following:

  * Pneumonia Severity Index (PSI) > 130 (Fine class V)
  * Patient placed on mechanical ventilation (invasive or not) for acute respiratory failure, with a PEEP level of 5 cm of water or more
  * Patient treated by high-flow oxygen therapy with a FiO2 of 50% or more and a P/F ratio less than 300
  * Patient treated by oxygen therapy with a partial rebreathing-mask with a reservoir bag, provided that the PaO2 is less than (cf. table):

Oxygen flow (L/min) 6 7 8 9 10 or more PaO2 (mmHg) less than 180 210 240 270 300

* Patient already treated by antibiotics (at least one dose since admission to hospital)
* Informed consent signed by the patient, its relatives or emergency procedure

On the sub-group of patients included with COVID19 :

* Diagnosis of COVID19 either as certain (PCR) or probable (evocative clinical and radiological features AND epidemic context AND absence of other microbiological documentation).
* Study drug infusion initiated no longer than 24 hours post first severity criterion ; in case of transfer from another hospital, this period will be prolonged to 48 hours
* Patient receiving the best available treatment as define by up-to-date scientific knowledge

Exclusion Criteria:

* Patient treated by vasopressors for septic shock at the time of inclusion
* Clinical history suggesting of aspiration of gastric content
* Patient treated by invasive mechanical ventilation within 14 days before current hospital admission
* Patient treated by antibiotics for a respiratory infection for more than seven days at the admission to the hospital (except if a pathogen resistant to this antibiotics is isolated)
* History of cystic fibrosis
* Post-obstructive pneumonia
* Patients in which rapid PCR-test is positive for flu
* Active tuberculosis or fungal infection
* Active viral hepatitis or active infection with herpes viruses
* Myelosuppression
* Decision of withholding mechanical ventilation or endotracheal intubation
* Hypersensitivity to corticosteroids
* Patient needing anti-inflammatory corticosteroids or substitutive hydrocortisone for any reason
* Patients under treatment by more than 15 mg/d of prednisone (or equivalent) for more than 30 days
* Patient already enrolled in another drug trial with mortality as an end-point. If the patient is already participating in another therapeutic trial with a different endpoint, the investigator must verify that inclusion in CAPE COD can not prejudice it.
* Pregnant or breastfeeding woman
* Patient on judicial protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 952 (Actual)
Dates: Start 2015-10-28 (Actual); Primary Completion 2020-07-19 (Actual); Study Completion 2020-08-28 (Actual)

PRIMARY OUTCOMES:
Day 28 all causes mortality | at day 28
Day 21 failure | at day 21
  For the sub-group of patients included with COVID19, failure is defined as death or need of respiratory support (mechanical ventilation or high-flow oxygen therapy);

SECONDARY OUTCOMES:
In patients non-invasively ventilated at inclusion, proportion of patients needing endotracheal intubation | Participants will be followed for the duration of hospital stay, for a maximum of 28 days
In patients non-ventilated at inclusion, proportion of patients requiring non-invasive ventilation | Participants will be followed for the duration of hospital stay, for a maximum of 28 days
In patients non-ventilated at inclusion, proportion of patients needing endotracheal intubation | Participants will be followed for the duration of hospital stay, for a maximum of 28 days
Day 28 ventilator-free-days | between 0 and day 28
Number of patients with vasopressor therapy initiation from inclusion to day 28 | between 0 and day 28
Day 28 vasopressor-free-days | between 0 and day 28
ICU and/or intermediate care unit LOS | Participants will be followed for the duration of hospital stay, for a maximum of 28 days
All-causes mortality at day 90 | at day 90
SF-36 Health Survey at day 90 | at day 90
Biomarkers: procalcitonin at baseline, day 3 and day 7 | at inclusion, day 3 and day 7
Biomarkers: C-reactive protein at baseline, day 3 and day 7 | at inclusion, day 3 and day 7
Biomarkers: plasmatic concentration of pro-inflammatory cytokines (IL-6, IL-20, IL-22, IL-22BP, HBD2, TNF) at baseline, day 3 and day 7 | at inclusion, day 3 and day 7
P/F ratio measured daily from baseline to day 7, at the end of treatment, at the end of ICU-stay and/or day 28 | measured daily from baseline to day 7, at the end of treatment i.e 14 days after the start of treatment, at the end of ICU-stay (for a maximum of 28 days) and/or day 28
SOFA calculated daily from baseline to day 7, at the end of treatment, at the end of ICU-stay and/or day 28 | calculated daily from baseline to day 7, at the end of treatment (i.e 14 days after the start of treatment), at the end of ICU-stay (for a maximum of 28 days) and/or day 28
Proportion of patients experiencing secondary infection during their ICU-stay | Participants will be followed for the duration of hospital stay, for a maximum of 28 days
Proportion of patients experiencing gastrointestinal bleeding during their ICU-stay | Participants will be followed for the duration of hospital stay, for a maximum of 28 days
Daily amount of insulin administered to the patient from day 1 to day 7 | Patients will be followed from day 1 to day 7
Weight-gain at baseline and day 7 | Patients will be followed at baseline and day 7

OTHER OUTCOMES:
P/F ratio measured daily from Day1 to Day7, at Day 14 and at Day 21 and/or at the end of ICU-stay | from day 1 to day 7, at day 14 and day 21 and/or at the end of ICU-stay
  Sub-group of patients included with COVID19
Proportion of patients needing endotracheal intubation | at day 21
  Sub-group of patients included with COVID19
Proportion of patients experiencing secondary infection during their ICU-stay | From baseline to day 21
  Sub-group of patients included with COVID19

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-François DEQUIN, MD-PhD, Principal Investigator — CHRU de TOURS
Locations (32):
- France (32):
  - Service de Réanimation - Unité de Soins Continus, CH d'Angoulême, Angoulême
  - Service de Réanimation Polyvalente, CH d'Argenteuil, Argenteuil
  - Service de Réanimation, CHR Metz-Thionville, Ars-Laquenexy
  - Service de Réanimation, Aulnay-sous-Bois
  - Service de Réanimation, Belfort
  - Service de Réanimation, Bourg-en-Bresse
  - Service de Réanimation HIA Clermont-Tonnerre, Brest
  - Service de Réanimation Médicale, CHU de Brest, Brest
  - Service de Réanimation, CHU Côte de Nacre, Caen
  - Service de Réanimation Médicale, Hôpital Louis Pasteur, Chartres, Chartres
  - Service de Réanimation Médicale Polyvalente, Hôpital G Montpied, Clermont-Ferrand
  - Service de Réanimation, Hôpital Louis Mourier, Colombes
  - Service de Réanimation Médicale, CHU de Dijon, Dijon
  - Service de Réanimation Médico-Chirurgicale, Hôpital Raymond Poincarré, APHP, Garches
  - Service de Réanimation Médicale, CHU de Grenoble, Grenoble
  - Service de Réanimation Polyvalente, CHD La Roche sur Yon, La Roche-sur-Yon
  - Service de Réanimation, CH Le Mans, Le Mans
  - Service de Réanimation Polyvalente, Hôpital Salengro, CHU de Lille, Lille
  - Service de Réanimation Polyvalente, CHU de Limoges, Limoges
  - Service de Réanimation Médicale, Hôpital Nord, Marseille
  - Service de Réanimation Polyvalente - Surveillance Continue, CH de Montauban, Montauban
  - Service de Réanimation Médicale, CHU de Nancy, Nancy
  - Service de Réanimation Polyvalente, Hôpital Hôtel Dieu, CHU de Nantes, Nantes
  - Service de Réanimation Médicale, CHR d'Orléans, Orléans
  - Service de Réanimation Médicale, Hôpital Cochin, APHP, Paris
  - Service de Réanimation et USC médico-chirurgicale, Hôpital Tenon, APHP, Paris
  - Service de Réanimation Médicale et Médecine Interne, CHU de Poitiers, Poitiers
  - Service des Maladies Infectieuses et Réanimation Médicale, CHU de Rennes, Rennes
  - Service de Réanimation, Saint-Brieuc
  - Service de Réanimation Polyvalente, CH de Saint Malo, St-Malo
  - Service de Réanimation Médicale, Nouvel Hôpital Civil, CHU de Strasbourg, Strasbourg
  - Service de Réanimation Médicale, Hôpital de Hautepierre, CHU de Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dequin PF, Heming N, Meziani F, Plantefeve G, Voiriot G, Badie J, Francois B, Aubron C, Ricard JD, Ehrmann S, Jouan Y, Guillon A, Leclerc M, Coffre C, Bourgoin H, Lengelle C, Caille-Fenerol C, Tavernier E, Zohar S, Giraudeau B, Annane D, Le Gouge A; CAPE COVID Trial Group and the CRICS-TriGGERSep Network. Effect of Hydrocortisone on 21-Day Mortality or Respiratory Support Among Critically Ill Patients With COVID-19: A Randomized Clinical Trial. JAMA. 2020 Oct 6;324(13):1298-1306. doi: 10.1001/jama.2020.16761. PMID 32876689
- [Derived] Friedrich JO, Gouvea Bogossian E. Hydrocortisone in Severe Community-Acquired Pneumonia. N Engl J Med. 2023 Aug 17;389(7):670-671. doi: 10.1056/NEJMc2307400. No abstract available. PMID 37585638
- [Derived] Dequin PF, Meziani F, Quenot JP, Kamel T, Ricard JD, Badie J, Reignier J, Heming N, Plantefeve G, Souweine B, Voiriot G, Colin G, Frat JP, Mira JP, Barbarot N, Francois B, Louis G, Gibot S, Guitton C, Giacardi C, Hraiech S, Vimeux S, L'Her E, Faure H, Herbrecht JE, Bouisse C, Joret A, Terzi N, Gacouin A, Quentin C, Jourdain M, Leclerc M, Coffre C, Bourgoin H, Lengelle C, Caille-Fenerol C, Giraudeau B, Le Gouge A; CRICS-TriGGERSep Network. Hydrocortisone in Severe Community-Acquired Pneumonia. N Engl J Med. 2023 May 25;388(21):1931-1941. doi: 10.1056/NEJMoa2215145. Epub 2023 Mar 21. PMID 36942789

DOCUMENTS (1):
  • Statistical Analysis Plan (2020-03-30): https://cdn.clinicaltrials.gov/large-docs/89/NCT02517489/SAP_000.pdf